CLINICAL TRIAL: NCT01558518
Title: Handheld Echocardiography in Clinical Practice
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Patricia A. Pellikka, MD, Professor of Medicine, Mayo Clinic
Other Study IDs: 11-008019
Record Dates: First submitted 2012-03-17; First posted 2012-03-20 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Cardiovascular Disease
Keywords: Handheld echocardiography; V-scan; Handheld ultrasound; Portable ultrasound
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Transthoracic echocardiography (TTE) represents an established and fundamental tool for the evaluation of patients with known or suspected cardiovascular disease. Recently, manufacturers have developed handheld echocardiograms small enough to fit in the pocket of a physician's lab coat. Studies assessing these handheld devices have several limitations. While they have generally evaluated the handheld devices favorably, previous studies has not consistently studied handheld devices under the best possible clinical conditions and have not necessarily highlighted the devices' limitations.

In this proposal, we seek to analyze the applicability of handheld echocardiograms to standard clinical practice. The investigators plan to use trained sonographers to perform handheld examinations on patients referred for TTE without established cardiovascular disease. The handheld images will be interpreted by experienced, consultant-level echocardiographers. The investigators then plan to compare findings from the handheld echocardiogram to the patient's standard clinical TTE.

ELIGIBILITY:
Inclusion criteria

* Adult patients referred for a resting transthoracic echocardiogram.

Exclusion criteria

* Referral for quantitative assessment of valvular heart disease
* Referral for strain imaging
* Referral for measurement of left atrial mechanical function or cardiac resynchronization studies
* Known diagnosis of congenital heart disease, restrictive cardiomyopathy, constrictive pericardial disease, or pulmonary hypertension
* Patients who have received left ventricular assist devices or those who have undergone cardiac transplants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Mayo Clinic Echocardiography Laboratory
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Pellikka, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Cullen MW, Blauwet LA, Vatury OM, Mulvagh SL, Behrenbeck TR, Scott CG, Pellikka PA. Diagnostic capability of comprehensive handheld vs transthoracic echocardiography. Mayo Clin Proc. 2014 Jun;89(6):790-8. doi: 10.1016/j.mayocp.2013.12.016. Epub 2014 Mar 29. PMID 24684783